CLINICAL TRIAL: NCT00097409
Title: A Phase II, Open-Label Study of Ispinesib in Subjects With Platinum/Taxane-Refractory or Resistant Relapsed Ovarian Cancer
Brief Title: Ispinesib In Subjects With Platinum-Taxane-Refractory Or Resistant Relapsed Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KSP20008
Record Dates: First submitted 2004-11-23; First posted 2004-11-24 (Estimated); Last update posted 2010-10-04 (Estimated); Status verified 2010-10

CONDITIONS: Ovarian Cancer
Keywords: ovarian cancer; platinum/taxane-refractory chemotherapy; Persistent; Recurrent
MeSH Terms: conditions — Ovarian Neoplasms; Recurrence | interventions — ispinesib

INTERVENTIONS:
Drug: Ispinesib

SUMMARY:
The purpose of this study is to determine how effective and safe a new investigational drug is in treating persistent or recurrent ovarian cancer in patients who have received a platinum/taxane based chemotherapy and whose disease continues to progress. The treatment involves a 1-hour treatment given intravenously (IV), and repeated once every 21 days. A patient may continue to receive the treatment as long as they are benefiting from the treatment. Blood samples will be taken at specific times over a 24 hour period to measure the amount of drug in your body at specific times after the drug is given. Blood samples will also be taken for routine lab tests such as complete blood counts and clinical chemistries. Physical exams will be performed before each treatment.

ELIGIBILITY:
Inclusion criteria:

* Must have a screening CA-125 of greater than or equal to 40 U/ml.
* Must have received only one prior platinum/taxane-based chemotherapy regimen.
* Blood tests will be done to check if blood counts are adequate for taking part in the study.

Exclusion criteria:

* Received more than 1 chemotherapy regimen in the past or have less than adequate liver and kidney function.
* Females who are pregnant or nursing.
* Any unstable, pre-existing major medical condition or history of other cancers.
* Have received an investigational drug, chemotherapy, radiation treatment or surgery within 28 days prior to entering the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2004-12; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Overall response rate of Ispinesib administered as a 1-hour intravenous infusion once every 21 days | once every 21 days

SECONDARY OUTCOMES:
Assess safety/tolerability, progression-free survival, time-to-response, response duration, and characteristics of Ispinesib administered as an infusion once every 21 days | once every 21 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (9):
- United States (9):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, New Orleans, Louisiana
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Mayfield Heights, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Abington, Pennsylvania
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Seattle, Washington
  - GSK Investigational Site, Madison, Wisconsin